CLINICAL TRIAL: NCT00333021
Title: Clinical Evaluation of GSK576428 (Fondaparinux Sodium) in Prevention of Venous Thromboembolism (VTE) After Abdominal Surgery
Brief Title: Abdominal Surgery Study Of GSK576428 (Fondaparinux Sodium)In Japanese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AR3106116
Record Dates: First submitted 2006-06-01; First posted 2006-06-02 (Estimated); Last update posted 2009-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Venous Thromboembolism
Keywords: Fondaparinux Abdominal surgery Japanese VTE
MeSH Terms: conditions — Venous Thromboembolism | interventions — Fondaparinux

INTERVENTIONS:
Drug: Fondaparinux sodium
Drug: GSK576428
  Other Names: Fondaparinux sodium

SUMMARY:
This study is phase 3 study for prevention of VTE in patients with abdominal surgery.

ELIGIBILITY:
Inclusion criteria:

* Patients aged >=40 years undergoing the following abdominal (diaphragm to pelvic floor) surgery under general anesthesia lasting more than 45 minutes.
* General or urologic surgery
* Cancer surgery
* Gynecologic surgery
* Radical surgery for pelvic malignancy

Exclusion criteria:

* Active, clinically significant bleeding Thrombocytopenia Body weight <40kg

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2006-05; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Venous thromboembolism and Major bleeding | Throughout entire study

SECONDARY OUTCOMES:
Incidence of Pulmonary embolism Incidence of Deep vein thrombosis Incidence of symptomatic Venous thromboembolism | Throughout entire study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (10):
- Japan (10):
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Nara
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo